CLINICAL TRIAL: NCT00015574
Title: Air Pollution and Implantable Cardioverter Defibrillators
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Tufts Medical Center (Other)
Other Study IDs: 9825-CP-002
Record Dates: First submitted 2001-04-20; First posted 2001-04-23 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Arrythmias
Keywords: arrhythmia; cardiac; air pollution; time series
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Community based studies have shown increased cardiovascular mortality associated with acute exposures to particulate air pollution. Electrocardiographic changes have also been reported in animals exposed to particles in controlled conditions. We have hypothesized that cardiovascular patients may experience life-threatening arrhythmias associated with particulate air pollution episodes. Implanted cardioverter defibrillator (ICD) devices continuously monitor the heart rhythm, and on detecting arrhythmias can initiate interventions. These devices provide a passive, continuous monitor of cardiac arrhythmias. We are assessing the association between community exposures to air pollution measured by ambient monitors and these cardiac arrhythmias detected by implanted cardioverter defibrillator devices.

DETAILED DESCRIPTION:
Records of cardiac arrhythmias detected in patients with implanted cardioverter defibrillators will be linked with measurements of the concentration and constituents of ambient particulate air pollution. Time series methods will be used to assess temporal associations, adjusting for seasonal, weekly, and diurnal patterns, meteorology, and co-pollutants. Characteristics of subjects showing the strongest air pollution associations will be assessed, as well as effect modification by medication and co-morbidities.

ICD patients are followed up clinically every three to six months. The ICD device is interrogated and data are retrieved by non-invasive radio frequency retrieval from the implanted device. Device performance is checked. Detected arrhythmias and therapeutic interventions are listed. For each detected episode, date and time is recorded, along with a short electrogram of the heartbeats immediately before and during the event.

Daily ambient particle mass (PM10 and PM2.5) and particle constituents have been measured in Boston since January 1995. The Massachusetts Department of Environmental Protection has measured concentrations of gaseous pollutants including carbon monoxide, nitrogen dioxide, ozone, and sulfur dioxide. Meteorological factors including temperature, humidity, and barometric pressure have been measured at the National Weather Service station at Logan airport. Meteorologic factors and gaseous co-pollutants will be considered as independent predictors of arrhythmic events, and as confounders of the particulate air pollution associations.

ELIGIBILITY:
The sample population consists of cardiac patients with implanted cardioverter defibrillator devices attending device clinics at the New England Medical Center (NEMC) Cardiac Electrophysiology and Pacemaker Laboratory. All patients with implanted ICD devices with event time and date recording living in the greater Boston area will be included.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 1998-09; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dockery, ScD, Study Director — Harvard School of Public Health (HSPH)
Locations (1):
- New England Medical Center, Cardiac Arrhythmia Service, Boston, Massachusetts, United States

REFERENCES:
- [Background] Peters A, Liu E, Verrier RL, Schwartz J, Gold DR, Mittleman M, Baliff J, Oh JA, Allen G, Monahan K, Dockery DW. Air pollution and incidence of cardiac arrhythmia. Epidemiology. 2000 Jan;11(1):11-7. doi: 10.1097/00001648-200001000-00005. PMID 10615837